CLINICAL TRIAL: NCT04504409
Title: Comparison of Efficacy of Dry Needling and Kinesio-taping on Myofascial Trigger Points in Patients With Common Shoulder Disorders
Brief Title: Comparison of Efficacy of Dry Needling and Kinesio-taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rüstem Mustafaoğlu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 127
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Myofascial Pain Syndromes
Keywords: shoulder pain; myofascial trigger point; dry needling; kinesio tape; exercise
MeSH Terms: conditions — Myofascial Pain Syndromes; Shoulder Pain; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (ExG) (Active Comparator): The exercise program consisted of; Codman , wand, stretching and strengthening exercises [25] applied twice a day, 5 times a week and duration of 3 weeks in all groups. All exercises were performed for 10 repetitions and 3 sets. Patients performed exercises with under supervision of physiotherapist in the clinic settings. In ExG, patients received only this exercise protocol for 3-weeks.
  Interventions: Other: Rehabilitation
- KT application combined with exercise (KTG) (Experimental): Before KT application, their skin was shaved, cleaned with alcohol, and dried. Prior to application, the patient was seated and asked to flex their neck laterally to the contralateral side and to rotate their head to the same side. KTs (Ares®) tape was used. The first strip was a Y-strip representative of the supraspinatus, which was applied from its insertion to origin with paper off tension. A Y-strip refers to a section of tape that has a portion cut down the middle to produce 2 tails. In KTG, patients wore the KT for a 3-week duration (renewed twice a week periodically in this time).
  Interventions: Other: Rehabilitation
- DN combined with exercise (DNG) (Active Comparator): The MTrP dry needling procedure employed was similar to the MTrP injection described by Hong. The MTrP was located by palpating the taut band and identifying the point of maximal tenderness. This was then firmly compressed by the index finger or middle finger of the nondominant hand to direct the placement of the needle tip while inserting the needle. The needle was inserted into the skin at a point above the taut band, approximately 1 cm from the MTrP region. After penetration of the needle into the subcutaneous layer, it was kept there and obliquely (about 45 degrees) directed to the MTrP region under the fingertip of the non-dominant hand. Then, the needle was inserted rapidly into the MTrP region and withdrawn rapidly. In DNG, patients received DN for a 3-week duration (twice a week periodically in this time).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Training

SUMMARY:
The aim of the current study was to investigate the effects of KT and DN combined with exercise on pain, range of motion (ROM), and upper extremity function in patients with common shoulder disorders.

DETAILED DESCRIPTION:
Shoulder pain is a common musculoskeletal problem seen in working population. The main contributor to nontraumatic upper-limb pain, in which chronicity and recurrence of symptoms are common. A common cause of muscle pain is myofascial pain caused by myofascial trigger points (MTrPs). Travel and Simons have described trigger points as 'a tender point on palpation characterized by referring pain, motor dysfunction and autonomic symptoms and usually located in the taut band or the fascia of the muscle. MTrPs in the shoulder muscles produce symptoms similar to those of other shoulder pain syndromes, including pain at rest and with movement, sleep disturbances and pain provocation during impingement tests. MTrPs are classified into active and latent trigger points. An active MTrP causes a clinical pain complaint. It is always tender, prevents full lengthening of the muscle, weakens the muscle, refers a patient-recognized pain on compression, mediates a local twitch response of muscle fibers when adequately stimulated and, when compressed within the patient's pain tolerance, produces referred motor phenomena and often autonomic phenomena, generally in its pain reference zone, and causes tenderness in the pain reference zone. A latent MTrP is clinically quiescent with respect to spontaneous pain; it is painful only when palpated. A latent MTrP may have all the other clinical characteristics of an active MTrP and always has a taut band that increases muscle tension and restricts range of motion. An alternative approach to the management of persons with shoulder problems consists of a treatment aimed at inactivating MTrPs and eliminating factors that perpetuate them. Manual techniques (such as compression on the trigger point or other massage techniques), cooling the skin with ethyl chloride spray and stretch and trigger point needling can inactivate MTrPs. MTrP inactivation may be combined with active exercises, postural correction, extracorporeal shock wave therapy, kinesio taping and relaxation if and when appropriate. Kinesio taping (KT) and dry needling (DN) are two common applications being used in treatment of acute and chronic musculoskeletal problems in recent years. Several therapies have been proposed for MTrPs, including KT, a relatively new method that has become widely used as a therapeutic tool in a variety of prevention and rehabilitation protocols. KT is an elastic cotton adhesive tape which is latex-free and can be used on any joint or muscle. Te exact mechanism by which KT functions remain unknown, though it is thought that its effectiveness may be mediated by cutaneous mechanoreceptors which would provide sensorimotor and proprioceptive feedback, and/or by mechanical restraint and inhibitory and excitatory nociceptive stimuli [16]. Various groups have shown that the use of KT can be beneficial, for example, by decreasing pain or by increasing range of motion (ROM) in shoulder pathologies. Among the non-pharmacological options, DN, despite the controversy, is currently considered one of the most effective interventions for the direct inactivation of MTrPs and is gaining attention for the treatment of MTrPs in musculoskeletal pain by targeting trigger points and non- trigger point structures. It is a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying trigger points, muscular and connective tissues without the use of injectate. A systematic review with meta-analysis reported that DN, compared with sham/placebo, can decrease pain immediately after treatment and in four weeks among patients with upper quarter myofascial pain syndrome. Another systematic review with metaanalysis reported that DN can be recommended to relieve MTrP pain of neck and shoulders in short and medium terms, but wet needling is more effective than DN in reducing MTrP pain in neck and shoulders in medium term.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they had unilateral non-traumatic shoulder pain (described as pain felt in the shoulder or upper arm) for at least six months, were between ages 18-60 years, and diagnosed with at least one active MTrP in shoulder region.

Exclusion Criteria:

* Patients who have been diagnosed with shoulder instability, shoulder fractures, neurological diseases, or other severe medical or psychiatric disorders will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3-weeks
  Pain intensity was assessed using the Visual Analog Scale (VAS), in which the patient is asked to indicate his/her perceived pain during rest, activity and at night (0-10 VAS, with 0 as no pain and 10 as worst imaginable pain.
Range of Motion | 3-weeks
  Limited and painful ROM is often observed in patients with shoulder disorders. Shoulder active ROM was measured in a supine position using a universal goniometer. The goniometer is a reliable instrument for measuring shoulder ROM . All measurements will be taken with patients standing. In this study, three repetitions were performed in each direction, and the average of three trials will determine the mean ROM values for each condition.

SECONDARY OUTCOMES:
Upper extremity functions | 3-weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item scale of disability symptoms used to assess a patient's health status. The scores obtained from all items are then used to calculate a score ranging from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Rüstem Mustafaoğlu, Principal Investigator — İstanbul Üniversitesi, Sağlık Bilimleri Fakültesi
Locations (1):
- Rüstem Mustafaoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roquelaure Y, Ha C, Leclerc A, Touranchet A, Sauteron M, Melchior M, Imbernon E, Goldberg M. Epidemiologic surveillance of upper-extremity musculoskeletal disorders in the working population. Arthritis Rheum. 2006 Oct 15;55(5):765-78. doi: 10.1002/art.22222. PMID 17013824
- [Result] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Result] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Alonso-Blanco C, Ge HY, Arendt-Nielsen L, Arroyo-Morales M. Muscle trigger points and pressure pain hyperalgesia in the shoulder muscles in patients with unilateral shoulder impingement: a blinded, controlled study. Exp Brain Res. 2010 May;202(4):915-25. doi: 10.1007/s00221-010-2196-4. Epub 2010 Feb 26. PMID 20186400
- [Result] Bron C, Dommerholt J, Stegenga B, Wensing M, Oostendorp RA. High prevalence of shoulder girdle muscles with myofascial trigger points in patients with shoulder pain. BMC Musculoskelet Disord. 2011 Jun 28;12:139. doi: 10.1186/1471-2474-12-139. PMID 21711512